CLINICAL TRIAL: NCT01103518
Title: Phase IV Study of the Use of Two Preparations of Ethinyl Estradiol and Cyproterone Acetate in Irregular Menstruation of Hyper-androgenic Origin
Brief Title: Ethinyl Estradiol and Cyproterone Acetate in Irregular Menstruation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundação Educacional Serra dos Órgãos (Other)
Responsible Party: Prof. Carlos Romualdo Barboza Gama, Fundação Educacional Serra dos Órgãos
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMI 1-16-08-09
Record Dates: First submitted 2010-04-12; First posted 2010-04-14 (Estimated); Last update posted 2010-08-06 (Estimated); Status verified 2010-04

CONDITIONS: Amenorrhea; Dysmenorrhea; Menstruation Disturbances; Hyperandrogenism
Keywords: Menstrual irregularity; Menstruation disturbances; Hyperandrogenism
MeSH Terms: conditions — Amenorrhea; Dysmenorrhea; Menstruation Disturbances; Hyperandrogenism | interventions — Cyproterone acetate, ethinyl estradiol drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination 1 (Experimental): Ethinyl Estradiol + Cyproterone acetate
  Interventions: Drug: Ethinyl Estradiol + Cyproterone acetate
- Combination 2 (Active Comparator): Ethinyl Estradiol + Cyproterone acetate
  Interventions: Drug: Ethinyl Estradiol + Cyproterone acetate

INTERVENTIONS:
Drug: Ethinyl Estradiol + Cyproterone acetate — Ethinyl Estradiol (0.035mg) + Cyproterone acetate (2mg), coated tablets. Each treatment cycle consists of one tablet, once per day for 21 days followed by a 7-day rest period. A total of 4 treatment cycles will be completed during the study treatment period.

SUMMARY:
This is a Phase IV, randomized, double-blind, comparative study of the use of two preparations of ethinyl estradiol and cyproterone acetate in the treatment of menstrual irregularities of hyper-androgenic origin.

ELIGIBILITY:
Inclusion Criteria:

* Female subject
* Premenopausal subject
* 18 years or older
* Medical history of irregular menses lasting at least 3 months
* Signature of informed consent

Exclusion Criteria:

* Pregnancy
* Use of hormonal contraceptives within 3 months of screening
* Primary bilateral oophorectomy
* Chemotherapy and / or radiotherapy within 6 months of screening
* Hysterectomy
* Myotonic dystrophy
* Galactosemia
* Galactorrhea
* History of tuberculosis or schistosomiasis
* Elevated prolactin / other significant laboratory alterations
* Diabetes
* Premature ovarian deficiency
* Sensitivity to any component of the drug formula

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-11 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Regular Menstruation | Treatment month 3
  Percentage of subjects with regular menstruation at the end of treatment month 3

SECONDARY OUTCOMES:
Menstrual flow | Treatment months 3
  Percentage of subjects with light, moderate, or heavy menstrual flow at treatment month 3
Menstrual colic | Treatment month 3
  Percentage of subjects reporting menstrual colic at pretreatment and at treatment month 3.
Global self evaluation scores | Treatment month 6
  Percentage of subjects with scores of 9 and 10 on the self evaluation of global condition.
Willingness to continue treatment | Treatment month 6
  Percentage of subjects willing to continue treatment with study drug
Safety | Treatment and follow-up period
  Incidence, duration and severity of adverse events, including laboratory tests.
Menstrual Flow | Treatment month 4
  Percentage of subjects with light, moderate, or heavy menstrual flow at treatment month 4
Menstrual Flow | Treatment month 5
  Percentage of subjects with light, moderate, or heavy menstrual flow at treatment month 5.
Menstrual Colic | Treatment month 4
  Percentage of subjects reporting menstrual colic at pretreatment and at treatment month 4.
Menstrual Colic | Treatment month 5
  Percentage of subjects reporting menstrual colic at pretreatment and at treatment month 5.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos RB Gama, M.D., Principal Investigator — Fundação Educacional Serra dos Órgãos; Carlos P Nunes, M.D., Study Director — Fundação Educacional Serra dos Órgãos
Locations (1):
- Hospital das Clínicas de Teresópolis, Teresópolis, Rio de Janeiro, Brazil